CLINICAL TRIAL: NCT07211490
Title: Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) in Pediatric Cerebellar Ataxia: A Randomized Controlled Trial
Brief Title: rTMS for Cerebellar Ataxia in Children
Acronym: rTMS CA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie Wan Yee Tso (Dr), Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rTMSCAHKU
Record Dates: First submitted 2025-10-02; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Cerebellar Ataxia
Keywords: TMS; Cerebellar ataxia; Children
MeSH Terms: conditions — Cerebellar Ataxia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional rTMS group (Experimental): The intervention group will receive 1 Hz rTMS for 15 minutes, followed by 1.5 hours of motor training.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS group (Sham Comparator): The sham group will not receive any Hz of rTMS for 20 minutes, followed by 1.5 hours of motor training.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — 1 Hz rTMS for 20 minutes, followed by 1.5 hours of motor training.
  Arms: Interventional rTMS group
Device: Sham Repetitive Transcranial Magnetic Stimulation — Sham Hz rTMS for 20 minutes, followed by 1.5 hours of motor training.
  Arms: Sham rTMS group

SUMMARY:
Dysfunction of the cerebellum can result in cerebellar ataxia (CA), typically marked by symptoms such as movement incoordination, gait instability, articulation disorder, oculomotor and swallowing difficulties. Children affected by paediatric cerebellar ataxia (PCA) often suffer from an array of motor symptoms, affecting their quality of life and psychosocial well-being. It was estimated that PCA affects 26/100,000 children worldwide for both genetic and acquired causes. Epidemiological data on PCA, however, are absent in the Hong Kong population.

PCAs comprise a varied group of cerebellar development disorders, marked by impaired balance and motor coordination (e.g., dysmetria and tremor) when performing voluntary movement. Clinical symptoms in children with PCA are related to lesioned localization - focal disorder of the cerebellar vermis leads to truncal instability, head titubation, and nystagmus; while lesioned cerebellar hemispheres results in ataxia gait (wide-staggering gait, tend to fall towards the affected side). These clinical symptoms result in functional difficulties involving balance and walking, reaching, grasping and manipulation, oculomotor and speech domains. Abnormalities of motor excitability have been reported in patients with cerebellar lesions - the motor threshold was found to be raised in the motor cortex contralateral to a hemi-cerebellar lesion.

With no effective pharmacological treatments available, rehabilitation serves as the primary treatment approach. Even though adaptive learning is affected by cerebellar lesion, motor learning is still possible via exercise interventions. Interventions may include compensatory (educate strategies to compensate for impairment) or restorative approaches (improve functions through training). While exercise interventions have been explored as a potential therapeutic approach for paediatric patients with cerebellar lesions or degeneration, the current evidence lacks robust, high-quality randomized controlled trials (RCTs) to substantiate their efficacy.

Existing evidence shows that cerebellar outputs project to several cortical areas, including the primary motor cortex (M1). CA patients with lesions in structures of the cerebellar efferent pathway exhibit reduced inhibition in the motor cortex. Selective modulation of the efferent pathways may offer an additional means of modulating cortical activity, thus improve motor coordination abilities in CA patients. With the development of non-invasive brain stimulation (NIBS) techniques, more research has been conducted using NIBS as treatment modalities for patients with CA. The most used NIBS techniques include repetitive transcranial magnetic stimulation (rTMS) and transcranial direct current stimulation (tDCS). Repetitive transcranial magnetic stimulation (rTMS) enables to modulate cortical excitability focally in conscious subjects; low-frequency stimulation (e.g., 1 Hz) is known to suppress cortical excitability, while higher frequencies (> 5 Hz) induce facilitation. These changes in excitability occur not only at the site of stimulation but also at other distant interconnected sites of a network. Both the excitatory stimulation and inhibitory stimulation approaches were adopted in existing adult studies. Paediatric patients with cerebellar lesions-caused by stroke, tumour, or genetic conditions-are thought to share the same pathophysiological basis as adults. Using contra-lesional inhibitory rTMS, França et al. demonstrated that the intervention is safe and feasible for adult patients with CA, showing a reduction in ataxic symptoms. Despite promising results in the adult population, it is still unclear whether rTMS can relieve ataxic symptoms and improve motor performance in children with CA.

To date, no studies have been published on the effects of rTMS on improving ataxic symptoms in children with cerebellar ataxia. However, emerging evidence suggests its potential utility. Using rTMS of 1 Hz to stimulate the cerebellar hemisphere ipsilateral to the ataxic side combined with mirror therapy, Cha et al. demonstrated that there was improvement in functional mobility as measured by 6-minute walk test and the timed up and go test. Supporting the feasibility of rTMS in paediatric motor rehabilitation, our pilot RCT (HKWC UW 23-492) found that contra-lesional inhibitory rTMS over M1 combined with motor training is safe and effective in improving motor performance in children with cerebral palsy. Comparative studies in older adults suggest that cerebellar rTMS was more effective than M1 rTMS for motor learning and the consolidation, likely due to the unique role of cerebellum in the integration and processing of multimodal sensory inputs to refine motor planning. These findings highlight the cerebellum as a promising neuromodulatory target for motor rehabilitation, warranting further investigation in paediatric cerebellar ataxia.

DETAILED DESCRIPTION:
To address the research gap, our study aims to use low frequency rTMS over the contra-lesional cerebellum in children with cerebellar ataxia. We aim to measure the reduction in ataxic symptoms, the improvement in motor performance functionally as well as using neuroimaging. We hypothesize that low frequency rTMS applied to the contra-lesional cerebellum will lead to reduced ataxic symptoms as measured by ataxia rating scales, improved motor abilities as measured by motor assessment scales, as well as showed improvement in structural as well as functional connectivity. Our study aims to use low frequency stimulation to the contra-lesional cerebellum which will be a safer option as no stimulation will be given to affected brain regions with abnormal brain changes or scarring. This study will be a prospective and randomized controlled study and aims to assess the treatment effect, and the sustainment of the treatment effect, of a 10-day treatment paradigm consisting of: 1) contra-lesional inhibitory rTMS and 2) post-treatment motor training in reducing ataxic symptoms in children with cerebellar ataxia. This study also aims to investigate the underlying neurophysiological mechanisms responsible for the rTMS treatment effect.

The specific hypotheses to be tested include:

* rTMS followed by motor training will reduce ataxic symptoms as reflected by ataxia rating scales (SARA and ICARS) to a greater extent than training alone in children with cerebellar ataxia.
* rTMS followed by motor training will lead to better quality of life (QoL) than training alone.
* rTMS followed by motor training will result in increased cortical plasticity compared to training alone.
* rTMS followed by motor training will result in brain microstructural changes demonstrated by DKI compared to training alone.
* rTMS followed by motor training will result in improvement in structural and functional connectivity demonstrated by DKI and resting state fMRI compared to training alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 4 years old - 18 years old fulfilling the following criteria: 1) diagnosis of cerebellar ataxia based on clinical history and neurological examination; 2) cerebellar lesion seen by MRI; 3) IQ ≥ 50 to ensure sufficient cognitive capacity for comprehending and adhering to motor training protocols.

Exclusion Criteria:

* Patients will be excluded if they have: 1) Sensory ataxia with etiologies involving the peripheral nerves or posterior columns of the spinal cord, 2) Any contra-indications to rTMS, 3) Severe spasticity (defined as a score of 4 in the Modified Ashworth Scale) and contractures, 4) Uncontrollable epilepsy defined as the occurrence of seizures despite the use of at least one anti-epileptic drug (AED) in adequate dose, 5) History of Botulinum toxin A injection or upper limb casting in previous 6 months, and 6) Cerebellar ataxia resulting from genetic conditions.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
The Scale for Assessment and Rating of Ataxia (SARA) | Day 10, 17 of intervention and 2 months post intervention.
  an evaluation tool for cerebellar ataxia patients. It consists of the following items: gait, stance, sitting, speech disturbance, finger chase, finger-nose test, fast alternating hand movements, and heel-shin slide.
The International Cooperative Ataxia Rating Scale (ICARS) | Day 10, 17 of intervention and 2 months post intervention.
  an assessment scale for severity of cerebellar ataxia. ICARS consists of 19 items divided into four sub-scores: posture and gait disturbances, (limb) kinetic functions, speech disorders, and oculomotor disorders.

SECONDARY OUTCOMES:
The 10 Metre Walk Test (10MWT) | Day 10, 17 of intervention and 2 months post intervention.
  an assessment with good reliability and validity to measure locomotor abilities in adults and children.
The Timed Up and Go Test (TUG) | Day 10, 17 of intervention and 2 months post intervention.
  a tool originally developed for frail adults/elderly to measure the time taken (in seconds) for an individual to rise from a chair, walk 3 meters, turns, walk back, and sit down. It is also proven that there are good psychometric properties to measure functional mobility in children and adolescents.
Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2), Subtests 4 and 7 | Day 10, 17 of intervention and 2 months post intervention.
  measure bilateral and upper limb coordination in children and adolescents aged between 4 and 21 years.
The Pediatric Balance Scale (PBS) | Day 10, 17 of intervention and 2 months post intervention.
  a measure of balance in school-age children, modified from Berg Balance Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No